CLINICAL TRIAL: NCT02400502
Title: Targeting Stress Reactivity in Schizophrenia: Integrating Coping Awareness Therapy (I-CAT) Pilot Trial
Brief Title: Integrated Coping and Awareness Training
Acronym: I-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1815; R21MH100250 (NIH)
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Treatment; Meditation; Mindfulness; Stress reactivity; First Episode Psychosis; Coping
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I-CAT Therapy (Experimental): Integrated Coping and Awareness Therapy is a six-month intervention designed to examine the physiological, biological, and psychological effects of meditation and mindfulness practice on individuals diagnosed with a psychotic disorder.
  Interventions: Behavioral: I-CAT Therapy

INTERVENTIONS:
Behavioral: I-CAT Therapy — I-CAT is a novel therapeutic intervention combining mindfulness and meditation strategies to improve stress reactivity and increase meaningful coping, as well as a range of possible proximal (e.g. autonomic, endocrine, immune indices of stress reactivity, symptom severity) and distal measures (function, relapse, quality of life). Participants meet weekly with a master's level clinician over the course of 20 weeks.

SUMMARY:
Integrated Coping and Awareness Therapy is a novel therapeutic intervention combining strategies to improve stress reactivity and increase meaningful coping, as well as a range of possible proximal (e.g. immune indices of stress reactivity, symptom severity) and distal measures (e.g. relapse, quality of life).

DETAILED DESCRIPTION:
Schizophrenia is one of the most devastating disorders that often results in a lack of functional recovery. Current treatments focused on remediating symptoms have shown only small successes in a return to functioning despite evidence of a dysregulated stress response. There is a fundamental gap in understanding the impact of allostatic overload in persons with schizophrenia that the investigators theorize is associated with deficits in functioning and with an increased vulnerability and relapse risk. The long-term goal is to test an intervention aimed at improving stress reactivity. The objective in this application is to develop and test the feasibility of a novel therapeutic intervention combining strategies to improve stress reactivity and increase meaningful coping. The central hypothesis is that an intervention that improves stress reactivity as measured proximally by endocrine, immune, and autonomic indices will result in improved adaptive capacity, better role functioning, reduced risk of relapse, and decreased likelihood of disability for people in the early stages of schizophrenia.

The rationale for the proposed research is that stress reactivity may be a modifiable risk factor underlying functional deficits in schizophrenia. The intervention integrates two treatment approaches. The first is based on research showing that mindfulness meditation practice is associated with alterations in the neural processing of stressful events and targets adaptive responses to stress. The second focuses on providing a buffer against stress by using the self-generation of adaptive emotions with a positive psychology intervention, which is potentially associated with building protective social resources. These complimentary interventions provide a comprehensive synergistic approach for this population that could lead to more adaptive coping responses and create a buffer against stress.

ELIGIBILITY:
Inclusion Criteria:

* Current or past diagnosis of a schizophrenia spectrum disorder.
* Has been receiving treatment for psychosis or taking medication for psychosis for less than 5 years.

Exclusion Criteria:

* Has been hospitalized in the last 3 months.
* Currently practicing meditation
* Current dependence on alcohol or drugs.
* History of significant neurological disorder.
* History of serious head injury (i.e., loss of consciousness longer than 15 minutes, no neuropsychological sequelae, no cognitive rehabilitation treatment post head injury).
* Illiteracy.
* Sensory limitation including visual (e.g., blindness, glaucoma, vision uncorrectable to 20/40) or hearing (e.g. hearing loss) impairments.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Salivary Cortisol at Six Months | Baseline, 6 Months
  Salivary cortisol measured before, during and after a social stressor test.

SECONDARY OUTCOMES:
Change from Baseline Urinary Oxidative Stress Level [Isoprostane] at Six Months | Baseline, 6 Months
Change from Baseline Positive and Negative Syndrome Scale (PANSS) Total Score at Six Months | Baseline, 6 Months
  The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 (no current symptomatology) to 210 (severely ill).
Change from Baseline Quality of Life Scale (QLS; Bilker et al., 2003) Total Score at Six Months | Baseline, 6 Months
  The Quality of Life Scale (QLS) is a semi-structured interview with 7-items that are rated on a 7-point scale with higher ratings reflecting less impaired functioning.
Change from Baseline Heart Rate Variability (HRV) Measurement at Six Months | Baseline, 6 Months
Change from Baseline Modified Differential Emotions Scale (mDES) Positive Emotion Sub Scale Score at Six Months | Baseline, 6 Months
  Rating scale that identifies strongest experiences of 20 emotions for the past week on a 5-point scale from (0 = not at all to 4= extremely). The mDES includes a Positive and Negative Emotion subscale.
Change from Baseline Perceived Stress Scale (PSS) Total Score at Six Months | Baseline, 6 Months
  The PSS is a 10-item, well validated and widely used self-report measure of the degree that situations in day-to-day life are perceived as stressful, unpredictable, uncontrollable, and how overloaded subjects find their lives. The 10 items are rated on a 5-point scale that ranges from 0 (never) to 4 (almost always). The PSS total score consists of the sum of the 10 PSS items and ranges from 0 (no subjective experience of stress) to 40 (overwhelmed with stress).
Change from Baseline Brief COPE Scale (Assisted Format) Total Score at Six Months | Baseline, 6 Months
  A short-version COPE Inventory. Assesses response to stress. 14 scales with two items each; self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion and self-blame. Reliability analyses exceeded alpha=0.60, except for venting, denial and acceptance, all of which exceed alpha = 0.50 (Carver et al 1997) Carver, C. S. (1997). International Journal of Behavioral Medicine, 4, 92-100
Change from Baseline Five Facet Mindfulness Questionnaire (FFMQ) Total Score at Six Months | Baseline, 6 Months
  The Five Facet Mindfulness Questionnaire (FFMQ) which assesses the five facets of being mindful in daily life: observing, describing, acting with awareness, non-reactivity to inner experience, and non- judging of inner experience. Each of the 39 items is rated using a Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true).
Change from Baseline Psychological Well-Being (PWB) Scale Total Score at Six Months | Baseline, 6 Months
  The Psychological Well-Being (PWB) Scale includes six sub scales (autonomy, environmental mastery, personal growth, purpose in life, positive relations with others, and self-acceptance) as well as a total score. The 54 items are rated on a 7-point Likert scale from 1 "strongly disagree" to 7 "strongly agree", with some items being reverse-scored.

CONTACTS AND LOCATIONS:
Overall Officials: Diana O Perkins, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; David L Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Piper Meyer-Kalos, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States